CLINICAL TRIAL: NCT06718205
Title: Open-label, Single-arm, Multicenter Phase II Study of Nimotuzumab Injection Combined With Sintilimab and Chemotherapy as First-line Treatment for Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Nimotuzumab Combined With Sintilimab and Chemotherapy for Advanced Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-Nim-ESCC-18
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — nimotuzumab; sintilimab; Cisplatin

STUDY DESIGN:
Intervention Model Description: nimotuzumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nimotuzumab (Experimental): Nimotuzumab+sindilimab+chemotherapy
  Interventions: Drug: Nimotuzumab; Drug: Sintilimab; Drug: Paclitaxel-albumin; Drug: Cisplatin

INTERVENTIONS:
Drug: Nimotuzumab — Combined chemotherapy phase Nimotuzumab 400mg，I.V.，D1，QW Maintenance treatment period:Until unbearable or PD Nimotuzumab 400mg，I.V.，D1，Q3W
Drug: Sintilimab — Sintilimab 200mg，I.V.，D1，Q3W，Until unbearable or PD
Drug: Paclitaxel-albumin — Paclitaxel-albumin 200 mg/m2，I.V.，D1，Q3W，4-6 Cycle
Drug: Cisplatin — Cisplatin:75 mg/m2，I.V.，D1,Q3W，4-6 Cycle

SUMMARY:
This study is a prospective, single-arm, multicenter study. The patients were given chemotherapy with nimotuzumab and sindilimab. To analyze the efficacy and safety of nimotuzumab combined with sindilizumab and chemotherapy in first-line treatment of advanced or recurrent or metastatic esophageal cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multicenter study. Patients with locally advanced, metastatic esophageal squamous cell carcinoma who had received previous (new adjuvant) / radical treatment (including radical surgical resection and radical chemoradiotherapy) who had relapsed more than 6 months and did not receive other antitumor treatment The patients were given 4-6 cycles of chemotherapy with nimotuzumab and sindilimab and TP (according to the degree of tolerance), and continued maintenance therapy with nimotuzumab and sindilimab. Medication continued until disease progression or the patient was intolerable or the patient died or withdrawal from the study, nimotuzumab and sindilimab for 2 years and follow-up observation for 1 year. To analyze the efficacy and safety of nytuzumab combined with cindilizumab and chemotherapy in first-line treatment of advanced or recurrent or metastatic esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

All of the following participants will be enrolled in this trial:

1. Patients voluntarily joined the study, signed informed consent, good compliance and follow-up.
2. unresectable locally advanced, unresectable recurrent or metastatic ESCC confirmed by histopathology (excluding mixed adenosquamous cell carcinoma type);
3. Patients who have not received previous systemic treatment, or have received previous (new) adjuvant treatment / radical treatment regimen (including radical surgical resection and radical chemoradiotherapy regimen) after recurrence for more than 6 months; Note: Including patients with reprogression after radiotherapy alone in late or recurrent non-target lesions. End of palliative treatment time to enrollment time of> 2 weeks for local lesions (non-target lesions);
4. Have at least one measured lesion according to the efficacy evaluation criteria of solid tumors version RECIST 1.1;
5. Male or female patients between the ages of 18 and 75;
6. Physical condition (PS) score of Eastern Oncology Cooperative Group (ECOG): 0-1;
7. The survival period is expected to exceed 3 months;
8. Having adequate organ and bone marrow function, that is, meeting the following criteria:

   A) Routine blood test criteria required (14, no blood transfusion and blood products within days, no correction with G-CSF and other hematopoietic stimulating factors):

   Hemoglobin content (HB): 100g / L; Leukocyte content (WBC) 3.0*10^9 / L; Neutrophil count (ANC) 1.5*10^9 / L; Platelet count (PLT) of 75*10^9 / L.

   B) Biochemical examination shall meet the following standards:

   Total serum bilirubin (TBIL) 1.5 times the upper limit of normal (ULN); ALT and AST≤2.5ULN; ALT and LT AST 5 ULN; Cr≤1.5ULN Or creatinine clearance (CCr) 60 ml/min; (Cockcroft-Gault formula) C) Full coagulation function, defined as international normalized ratio (INR) or prothrombin time (PT) 1.5 times ULN; And d) Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) low normal value (50%); E) myocardial zymogram: within the normal range.
9. Women of childbearing age should take appropriate contraceptive measures from screening to 3 months after the cessation of study treatment, and they must be non-lactating patients. Before starting administration, the pregnancy test was negative or no risk of pregnancy was demonstrated by meeting one of the following criteria:

A) Postmenopause was defined as age greater than 50 years and amenorrhea for at least 12 months after cessation of all exogenous hormone replacement therapy; B) Women younger than 50 years old can also be considered postmenopausal if amenorrhea for 12 months or more after stopping all exogenous hormone therapy, and luteinizing hormone (LH) and follicular stimulating hormone (FSH) levels are within the range of laboratory postmenopausal reference values; And c) had ever undergone irreversible sterilization procedures, including hysterectomy, bilateral oophorectomy or bilateral tubal resection, except for bilateral tubal ligation. For men, give consent to appropriate contraception or surgical sterilization during the trial and 8 weeks after the last dose of trial drug;

Exclusion Criteria:

* 1) Patients who have previously received treatment with anti EGFR monoclonal antibodies or any anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibodies; 2) Esophageal squamous cell carcinoma that tends to be completely obstructed under endoscopy and requires interventional treatment to relieve obstruction; 3) Patients with high risk of bleeding or perforation due to obvious invasion of adjacent organs (large arteries or trachea) of esophageal lesions by tumors, or patients who have already formed fistulas; 4) Received major surgical treatment, open biopsy, or significant traumatic injury within 28 days prior to enrollment; 5) There are multiple factors that can affect the use of therapeutic drugs, such as inability to swallow or chronic diarrhea or intestinal obstruction, significant impact on drug administration and absorption, or a known history of severe allergies to any of the study drug ingredients.

  6) Patients who have received traditional Chinese medicine anti-tumor treatment within the past 2 weeks (including medicinal herbs such as brucea, coix seed, polysaccharides from shiitake mushrooms, cantharides, toad skin, astragalus, Sophora flavescens, Polygonatum sibiricum, and Hedyotis chinensis), but have been taking traditional Chinese medicine anti-tumor treatment for more than 2 weeks are allowed to be enrolled; 7) The burden of liver metastases accounts for over 50% of the entire liver volume; 8) Patients with any severe and/or uncontrolled illnesses, including:
  1. Patients with poor blood pressure control (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) using antihypertensive drugs; Or use two or more antihypertensive drugs to control blood pressure in patients; Patients who have previously experienced hypertensive crisis or hypertensive encephalopathy;
  2. Patients with grade I or above myocardial ischemia or infarction, arrhythmia (including QTc interval greater than 450ms in males and greater than 470ms in females), and ≥ grade 2 congestive heart failure (NYHA classification), severe/unstable angina pectoris, as well as those who have undergone coronary/peripheral artery bypass surgery;
  3. Active or uncontrolled severe infection (≥ CTCAE level 2 infection), known to have active pulmonary tuberculosis;
  4. Renal failure requires hemodialysis or peritoneal dialysis
  5. Liver diseases such as cirrhosis, decompensated liver disease, and chronic active hepatitis;
  6. Poor control of diabetes (FBG>10mmol/L);
  7. Urine routine shows urinary protein ≥++and confirms 24-hour urinary protein quantification>1.0 g; 9) Long term untreated wounds or fractures; 10) Known presence of symptomatic central nervous system metastases and/or cancerous meningitis; 11) Ascites with clinical significance, including any ascites that can be detected during physical examination, ascites that has been treated in the past or still requires treatment, and only those with imaging showing a small amount of ascites but no symptoms can be selected; 12) Patients with equal amounts of fluid accumulation in both pleural cavities, or a large amount of fluid accumulation in one pleural cavity, or those who have caused respiratory dysfunction and require drainage; 13) Suffering from interstitial lung disease that requires steroid hormone therapy; 14) Uncontrolled metabolic disorders or other non malignant tumor organs or systemic diseases or secondary reactions to cancer, which can lead to higher medical risks and/or uncertainty in survival evaluation; 15) Individuals with a history of abuse of psychotropic drugs who are unable to quit or have mental disorders; 16) Individuals with a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 17) History of other primary malignant tumors, except for the following:

  <!-- -->

  1. Complete remission of malignant tumors for at least 2 years prior to enrollment and no need for additional treatment during the study period;
  2. Non melanoma skin cancer or malignant freckle nevi that have been adequately treated and have no evidence of disease recurrence;
  3. In situ cancer with sufficient treatment and no evidence of disease recurrence; 18) There is any history of immune related illness or treatment that:

  <!-- -->

  1. Existence of any active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; subjects with asthma requiring bronchodilators for medical intervention cannot be included); However, the following patients are allowed to be included: vitiligo, psoriasis, alopecia without systemic treatment, well controlled type I diabetes, hypothyroidism with normal thyroid function after replacement treatment;
  2. Diagnosed with immunodeficiency or undergoing systemic glucocorticoid therapy or any other form of immunosuppressive therapy (prednisone or other therapeutic hormones at a dose>10mg/day), and continued to be used within 2 weeks prior to the first dose;
  3. Received any live vaccine, attenuated vaccine (including anti infective vaccines such as influenza vaccine, varicella vaccine, etc.) or inactivated vaccine within 4 weeks before enrollment, and planned to receive live vaccine/attenuated vaccine/inactivated vaccine during the study period; Used systemic immune stimulatory agents (including but not limited to interferon and IL-2) within 2 weeks prior to the start of the study treatment; 19) During pregnancy or lactation, 20) According to the researchers' judgment, there are accompanying diseases that pose a serious threat to patient safety or affect the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
PFS | about 2 years
  the first progression disease or death (whichever occurs first) from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Feng Wang, Zhengzhou, Henan, China